CLINICAL TRIAL: NCT02087488
Title: Auricular Acupuncture for Primary Insomnia
Acronym: AAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li ying, Principal Investigator, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011SZ0302-3
Record Dates: First submitted 2014-02-28; First posted 2014-03-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Primary Insomnia
Keywords: primary insomnia; auricular acupuncture
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture, Ear; Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- auricular acupuncture(AA) & Eszopiclone (Experimental): The disposable Seirin Pyonex Needle will be chosen as AA material to attach every 3 days for 4 weeks, meanwhile, oral Eszopiclone 1 piece (3mg) will be applied 15 minutes before going to sleep everyday for 4 weeks. The manufacturer of disposable Seirin Pyonex Needles is Seirin Corporation, a Japanese company.
  Interventions: Other: auricular acupuncture(AA); Drug: Eszopiclone
- placebo AA & Eszopiclone (Placebo Comparator): The disposable Pyonex Zero Needle, a non-invasive material will be chosen as placebo AA, with auricular acupoints have no certain effect on PI. Additionally, 1 piece (3mg) Eszopiclone will be administrated to participants 15 minutes before going to sleep everyday for 4 weeks.
  Interventions: Other: placebo AA; Drug: Eszopiclone

INTERVENTIONS:
Other: auricular acupuncture(AA) — Auricular acupoints: Shenmen (TF4), Heart (CO15), Subcortex (AT4), modifying points according to different patterns.
  Auricular attachment material: disposable Seirin Pyonex Needle Seirin Pyonex Needle manufacturer: Seirin Corporation, a Japanese company. Medical Device Certification number: No. 15500BZZ00806000.
  Treatment frequency: every 3 days.
  Duration: 4 weeks.
  Arms: auricular acupuncture(AA) & Eszopiclone
Other: placebo AA — Auricular acupoints: Wrist (SF1), Clavicle (SF6), Shoulder (SF4、5), Tooth (LO1), Tonsil (LO7, 8, 9).
  Auricular attachment material: the disposable Pyonex Zero Needle Pyonex Zero Needle manufacturer: Seirin Corporation, a Japanese company.
  Treatment frequency: every 3 days.
  Duration: 4 weeks.
  Arms: placebo AA & Eszopiclone
Drug: Eszopiclone — Dosage form: tablet.
  Dosage: 1 piece (3mg).
  Drug manufacturer: Kanghong pharmaceutical limited liability company, Chengdu.
  Production license: NO. H20100074 approved by the state.
  Treatment frequency: 15 mins before going to bed everyday.
  Duration: 4 weeks.
  Other Names: Lunesta or Estorra

SUMMARY:
This double-blind RCT will evaluate the therapeutic effectiveness and safety of auricular acupuncture(AA) for primary insomnia(PI) .

DETAILED DESCRIPTION:
Investigators will conduct a 2-year clinical trial on auricular acupuncture (AA) for primary insomnia (PI), which is a double-blind (patient-blind and assessor-blind) RCT. 288 patients will be randomly assigned into 2 groups: the treatment group (Group A) and the control group (Group B). Group A will be treated with AA plus oral Eszopiclone, while Group B will be treated with sham AA plus oral Eszopiclone. All patients will receive a continuous 4-week treatment and 28-week follow-up. The data will be analyzed by the third party who is not clear about allocation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of PI according to DSM-5;
* Aged 18-64 (including 18 and 64);
* Provided a signed written consent form.

Exclusion Criteria:

* The patient has somatic disease like severe respiratory, circulatory, endocrine system disease and hepatic/renal insufficiency;
* The patient suffers from moderate / major depression (BDI score ≧ 8 points), moderate / severe anxiety disorder (SAS score ≧ 61 points) or any other serious mental disease;
* The patient who abuse drug alcohol or substance;
* The patient suffers from dementia or any other severe cognitive impairment;
* The patient is in pregnancy or lactation period;
* Patient who is a night worker or stick to irregular sleep pattern, and can't or don't want to terminate this kind of work mode;
* The patient has history of suicide or suicidal tendency;
* The patient is allergic to Eszopiclone or any other sedative-hypnotic drugs;
* The patient who has taken psychiatric, hypnotic or antihistamine drugs during the last 4 weeks before baseline, however, the patient who use the prescription or nonprescription hypnotic drugs no more than twice a week can be recruited as soon as drug withdrawal;
* The patient who is receiving ongoing psychological treatment;
* The patient who has obstructive sleep apnea, restless leg syndrome, sleep rhythm disorders, parasomnias, etc.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sleep Onset Latency (SOL) | Change from baseline in SOL at 4 weeks
  SOL is one of the sleep parameters mainly measured by actigraphy and sleep diaries, referring to the time it takes to fall asleep, starting from the moment of having intention to fall asleep, stopping at the moment of getting a 5-minute continuous sleep.
Wake After Sleep Onset (WASO) | Change from baseline in WASO at 4 weeks
  WASO is one of the sleep parameters mainly measured by actigraphy and sleep diaries, referring to the total time of awakening which from the initial sleep onset to the last awakening.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index(PSQI) | Change from baseline in PSQI at 4 weeks
Insomnia Severity Index (ISI) | Change from baseline in ISI at 4 weeks
Beck Depression Inventory (BDI) | Change from baseline in BDI at 4 weeks
State-Trait Anxiety Inventory (STAI) | Change from baseline in STAI at 4 weeks
Self-rating Anxiety Scale (SAS) | Change from baseline in SAS at 4 weeks
The Epworth Sleeping Scale (ESS) | Change from baseline in ESS at 4 weeks
Flinders Fatigue Scale (FFS) | Change from baseline in FFS at 4 weeks
The MOS 36-Item Short-Form Health Survey questionnaire (SF-36) | Change from baseline in SF-36 at 4 weeks
Total Sleep Time (TST) | Change from baseline in TST at 4 weeks
  TST is one of the sleep parameters mainly measured by actigraphy and sleep diaries, referring to actually time slept, it's the amount of time from the initial sleep to final awakening, excluding the awake time.
Sleep Efficiency (SE) | Change from baseline in SE at 4 weeks
  SE is one of the sleep parameters mainly measured by actigraphy and sleep diaries, sleep efficiency percentage = [total sleep time/total time in bed] ×100%.
Number of awakenings (nWAK) | Change from baseline in nWAK at 4 weeks
  Obtained by actigraphy and sleep diaries, it's the number of awakening times from the initial sleep onset to the end of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Professor, Study Chair — Faculty of Acupuncture & Tuina，Chengdu University of Traditional Chinese Medicine; Xi Wu, A.P., Study Director — Faculty of Acupuncture & Tuina，Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu university of Traditonal Chinese Medcine, Chengdu, Sichuan, China